CLINICAL TRIAL: NCT02306694
Title: Prospective Biomarkers of Bone Metabolism in Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e11104
Record Dates: First submitted 2014-11-25; First posted 2014-12-03 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Hemophilia; Bone Disease
Keywords: hemophilia; bone disease; clinical study; biomarkers
MeSH Terms: conditions — Hemophilia A; Bone Diseases | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental): Everyone receives Advate (antihemophilic factor) on Day 1 and 3.
  Interventions: Drug: Advate

INTERVENTIONS:
Drug: Advate — Patients who are currently taking Advate as their factor replacement will be eligible for the 5-day study.
  Other Names: Antihemophilic Factor (Recombinant)

SUMMARY:
One of the major shortcomings in studying bone disease in hemophilia is the lack of fracture outcome data demonstrating the clinical significance of decreased BMD and altered bone biomarkers in the hemophilia population. This study demonstrates that PwH have an increased risk of fracture compared to the general population and that the issue of bone health will increase in importance as the PwH population ages.

DETAILED DESCRIPTION:
This is a pilot study to determine the impact of factor replacement on bone biomarkers in up to 20 hemophilia A subjects. Subjects will be recruited over 1 year for the 5-day protocol.

Following a 72-hour washout period, factor levels and bone biomarkers will be followed before and after 50 units/kg replacement on Day 1 and 20 units/kg replacement on Day 3. Each subject can serve as their Figure 4. Fracture rates in PwH compared to historic controls.

ELIGIBILITY:
Inclusion Criteria:

1. Males with a diagnosis of hemophilia A with a historic baseline FVIII level ≤ 2%.
2. Age > 16 years old
3. Currently using ADVATE as FVIII replacement therapy

Exclusion Criteria:

1. Subject or guardian is unwilling or unable to give written informed consent and/or assent
2. Joint or muscle bleeding within 2 weeks of Study Day 1
3. Presence of a current factor inhibitor (>0.6 BU/mL via Nijmegan-modified Bethesda assay)
4. Known collagen vascular bone disease.

Ages: 16 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Taylor, MD, PhD, Principal Investigator — Oregon Health and Science
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Plug I, Van Der Bom JG, Peters M, Mauser-Bunschoten EP, De Goede-Bolder A, Heijnen L, Smit C, Willemse J, Rosendaal FR. Mortality and causes of death in patients with hemophilia, 1992-2001: a prospective cohort study. J Thromb Haemost. 2006 Mar;4(3):510-6. doi: 10.1111/j.1538-7836.2006.01808.x. PMID 16460432
- [Background] Siboni SM, Mannucci PM, Gringeri A, Franchini M, Tagliaferri A, Ferretti M, Tradati FC, Santagostino E, von Mackensen S; Italian Association of Haemophilia Centres (AICE). Health status and quality of life of elderly persons with severe hemophilia born before the advent of modern replacement therapy. J Thromb Haemost. 2009 May;7(5):780-6. doi: 10.1111/j.1538-7836.2009.03318.x. Epub 2009 Feb 12. PMID 19220727
- [Background] Gerstner G, Damiano ML, Tom A, Worman C, Schultz W, Recht M, Stopeck AT. Prevalence and risk factors associated with decreased bone mineral density in patients with haemophilia. Haemophilia. 2009 Mar;15(2):559-65. doi: 10.1111/j.1365-2516.2008.01963.x. Epub 2009 Feb 1. PMID 19187193
- [Background] Wallny TA, Scholz DT, Oldenburg J, Nicolay C, Ezziddin S, Pennekamp PH, Stoffel-Wagner B, Kraft CN. Osteoporosis in haemophilia - an underestimated comorbidity? Haemophilia. 2007 Jan;13(1):79-84. doi: 10.1111/j.1365-2516.2006.01405.x. PMID 17212729
- [Background] Barnes C, Wong P, Egan B, Speller T, Cameron F, Jones G, Ekert H, Monagle P. Reduced bone density among children with severe hemophilia. Pediatrics. 2004 Aug;114(2):e177-81. doi: 10.1542/peds.114.2.e177. PMID 15286254
- [Background] Gallacher SJ, Deighan C, Wallace AM, Cowan RA, Fraser WD, Fenner JA, Lowe GD, Boyle IT. Association of severe haemophilia A with osteoporosis: a densitometric and biochemical study. Q J Med. 1994 Mar;87(3):181-6. PMID 8208906
- [Background] Tlacuilo-Parra A, Morales-Zambrano R, Tostado-Rabago N, Esparza-Flores MA, Lopez-Guido B, Orozco-Alcala J. Inactivity is a risk factor for low bone mineral density among haemophilic children. Br J Haematol. 2008 Mar;140(5):562-7. doi: 10.1111/j.1365-2141.2007.06972.x. PMID 18275434
- [Background] Amorosa V, Tebas P. Bone disease and HIV infection. Clin Infect Dis. 2006 Jan 1;42(1):108-14. doi: 10.1086/498511. Epub 2005 Nov 30. PMID 16323100
- [Background] Anagnostis P, Vakalopoulou S, Vyzantiadis TA, Charizopoulou M, Karras S, Goulis DG, Karagiannis A, Gerou S, Garipidou V. The clinical utility of bone turnover markers in the evaluation of bone disease in patients with haemophilia A and B. Haemophilia. 2014 Mar;20(2):268-75. doi: 10.1111/hae.12271. Epub 2013 Oct 7. PMID 24118364
- [Background] Liel MS, Greenberg DL, Recht M, Vanek C, Klein RF, Taylor JA. Decreased bone density and bone strength in a mouse model of severe factor VIII deficiency. Br J Haematol. 2012 Jul;158(1):140-3. doi: 10.1111/j.1365-2141.2012.09101.x. Epub 2012 Apr 2. No abstract available. PMID 22469061
- [Background] Kempton CL, Antun A, Antoniucci DM, Carpenter W, Ribeiro M, Stein S, Slovensky L, Elon L. Bone density in haemophilia: a single institutional cross-sectional study. Haemophilia. 2014 Jan;20(1):121-8. doi: 10.1111/hae.12240. Epub 2013 Aug 1. PMID 23902277
- [Background] Lee SK, Lorenzo J. Cytokines regulating osteoclast formation and function. Curr Opin Rheumatol. 2006 Jul;18(4):411-8. doi: 10.1097/01.bor.0000231911.42666.78. PMID 16763463
- [Background] Brinker MR, O'Connor DP. The incidence of fractures and dislocations referred for orthopaedic services in a capitated population. J Bone Joint Surg Am. 2004 Feb;86(2):290-7. PMID 14960673
- [Background] Roche AF, Roberts J, Hamill PV. Skeletal maturity of youths 12--17 years racial, geographic area, and socioeconomic differentials. United States, 1966-1970. Vital Health Stat 11. 1978 Oct;(167):1-98. No abstract available. PMID 214960

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label
Started | 16
Completed | 12
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
Weight [Mean (Standard Deviation); unit: lb] | 149.3 (192.9)

OUTCOME MEASURES:

1. Primary Outcome: Bone Biomarker Density (BMD)
Description: BMD was measured as Z-scores/T-scores using Dual-Energy X-ray Absorptiometry (DEXA) scanning; specifically looking at Spine, Hip/Neck, and Hip total scores. BMD Z-scores compare what would be expected in someone your age and body size. A Z-score, is a unit of standard deviation, where above 0 would indicate the bones are more dense than expected, while a Z-score below 0 would indicate the bones were less dense.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Open Label
Number analyzed (Participants) | 12
Z-Score
  Spine BMD (Spine L1-L4 Z-score) | -0.74 (1.22)
  Hip Total BMD | -0.16 (1.12)
  Hip Neck BMD | -0.16 (1.23)

2. Primary Outcome: Joint Health
Description: Hemophilia Joint Health Score (HJHS); with a higher score representing worst outcomes, scores could range from 0 (no problems) to a max score of 120 (severe problems).
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 12
score on a scale | 19.91 (16.26)

3. Primary Outcome: Quality of Life Using the VAS and EQ-5D-3L
Description: Visual Analog Scale (VAS) via the EQ-5D-3L was used to report participants self-rated health. EQ-5D-3L total score ranges from 5 (no problems) to 15 (significant problems). VAS scores could range from 0 (worst health ever) to 100 (best health ever).
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 12
score on a scale
  EQ-5D-3L | 6.92 (1.83)
  VAS | 82.42 (15.08)

4. Primary Outcome: Plasma Cytokine Concentration Differences From 0-hour to 24-hour
Description: cytokines were measured using ELISA/magnetic bead multiplex kits. We calculated concentration change from hour 0 to hour 24. Cytokines: FGF, C-Terminal telopeptide (CTX-1), Dickkopf WNT signaling pathway inhibitor 1(DKK1), Eotaxin, fibroblast growth factor 23(FGF23), interferon gamma, interleukin 13, interleukin 1 beta, interleukin receptor 1 antagonist, interleukin 2, interleukin 4, interleukin 6, interleukin 17, interleukin 8, interleukin 9 Insulin, interferon gamma induced protein 10 (IP10), Leptin, monocyte chemoattractant protein1, monocyte chemoattractant protein1, macrophage inflammatory protein 1a (MIP1a), osteoclasts, Osteoprotegerin, osteopontin, platelet derived growth factors, parathyroid horomone, Recepter activator of nuclear factor kappa-B ligand (RANKL), chemokine ligand 5, sclerostin, transforming growth factor-beta 1, transforming growth factor beta 2, transforming growth factor beta 3, tumor necrosis factor alpha, vascular endothelial growth factor, MIP1b.
Time Frame: 24 hours
Population: Some participant samples were unable to be analyzed at all time points due to poor sample quality or other factors.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Open Label
Number analyzed (Participants) | 12
pg/mL
  Basic FGF: number analyzed (Participants) | 4
  Basic FGF | 2.04 (1.78)
  C-Terminal telopeptide | 0.03 (0.12)
  DKK1 | -7.73 (15.63)
  Eotaxin | -2.84 (14.09)
  fibroblast growth factor 23: number analyzed (Participants) | 3
  fibroblast growth factor 23 | -6.72 (9.95)
  interferon gamma: number analyzed (Participants) | 7
  interferon gamma | 0.12 (0.52)
  interleukin 13: number analyzed (Participants) | 3
  interleukin 13 | -0.76 (1.52)
  Interleukin 1 beta: number analyzed (Participants) | 7
  Interleukin 1 beta | -0.12 (0.19)
  interleukin receptor 1 antagonist: number analyzed (Participants) | 11
  interleukin receptor 1 antagonist | -131.72 (429.93)
  interleukin 2: number analyzed (Participants) | 3
  interleukin 2 | 0.71 (1.16)
  interleukin 4: number analyzed (Participants) | 5
  interleukin 4 | -0.28 (0.39)
  interleukin 6: number analyzed (Participants) | 7
  interleukin 6 | 0.22 (0.38)
  interleukin 17: number analyzed (Participants) | 3
  interleukin 17 | -0.13 (0.80)
  interleukin 8: number analyzed (Participants) | 9
  interleukin 8 | -0.56 (0.99)
  interleukin 9: number analyzed (Participants) | 10
  interleukin 9 | -14.83 (14.03)
  Insulin | -279.39 (1518.67)
  IP10: number analyzed (Participants) | 10
  IP10 | -10.06 (36.49)
  Leptin | -208.39 (6728.25)
  MCP1: number analyzed (Participants) | 8
  MCP1 | -6.42 (7.53)
  MIP1a: number analyzed (Participants) | 7
  MIP1a | -0.23 (0.40)
  osteoclasts | -2146.62 (5921.06)
  osteoprotegerin: number analyzed (Participants) | 11
  osteoprotegerin | 113.70 (328.53)
  osteopontin | -493.87 (6795.35)
  platelet derived growth factors: number analyzed (Participants) | 3
  platelet derived growth factors | -103.83 (156.52)
  parathyroid horomone: number analyzed (Participants) | 11
  parathyroid horomone | -6.72 (25.70)
  RANKL | 228.10 (277.99)
  chemokine ligand 5 | -414.77 (681.82)
  sclerostin: number analyzed (Participants) | 6
  sclerostin | -398.13 (838.83)
  transforming growth factor-beta 1 | -519.05 (772.15)
  transforming growth factor beta - 2 | -10.08 (16.43)
  transforming growth factor beta - 3 | -0.74 (1.49)
  tumor necrosis factor alpha | -1.09 (2.76)
  VEGF | -4.03 (12.17)
  MIP1b | -7.19 (9.36)

5. Other Pre Specified Outcome: Medication Adherence
Description: VERITAS instrument self-reported compliance with factor replacement regimen. The VERITAS is composed of 6 subsections, where scores range from 1 (best adherence) to 5 (worst adherence). A total score was calculated with the minimum score of 24 (most adherent) and a maximum score of 120 (least adherent)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 12
score on a scale | 56.25 (5.29)

6. Other Pre Specified Outcome: Hemophilia Activities List (HAL) and the International Society of Thrombosis and Hemostasis- Bleeding Assessment Tool (ISTH-BAT)
Description: The HAL is used to assess physical activity; scores range from 42 (severe problems) to 252 (no problems). The ISTH-BAT was used to evaluate bleeding phenotype. Each section was scored using a 0 to 4 scale for each of the 12 subsections. A total score was calculated by taking the sum of each section, resulting in a range of scores from 0 (no bleeding history) to 48 (most extensive clinical intervention for bleeding)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 12
score on a scale
  HAL | 226 (41.78)
  ISTH-BAT | 16.92 (6.56)

7. Other Pre Specified Outcome: Participant Quality of Life
Description: Haem-A-QoL was used to assess various components indicating participants quality of life. Haem-A-QoL is composed of 10 subsections with 3-8 questions in each. Questions are rated from 1 to 5, with 5 being the most negative influence on quality of life. Some questions are worded in the inverse, such that the 1 corresponds to the greatest negative impact on quality of life. In this case, the score is inverted to match the remainder of questions for statistical analysis. A Transformed scores is calculated for each subsection and for the total of all the subjections. The scores range from 0 (best quality of life) to 225 (worst quality of life).
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 12
score on a scale | 113.83 (58.19)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02306694/Prot_SAP_000.pdf